CLINICAL TRIAL: NCT04675385
Title: Hyaluronic Acid 0.2% Application Enhanced Chronic Periodontitis Treatment in Non-surgical Phase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Thu Thuy, DDS, PhD, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1852/QD-DHYD
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Chronic Periodontitis, Hyaluronic Acid
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: Participants from 18 years old with a minimum number of 20 teeth who came for periodontitis treatment, were recruited at the Department of Periodontology, Faculty of Odonto-Stomalogy, the University of Medicine and Pharmacy at Ho Chi Minh City (FOS-UMPH.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: 0.2% hyaluronic acid gel — In this split mouth study, 733 periodontal pockets of 28 patients with moderate to severe chronic periodontitis were chosen for investigation. They were divided into 2 groups: control group and experimental group. The experimental group received sub-gingival administration of 1 ml of 0.2% hyaluronic acid gel into each pocket immediately after root planing and then after 1 week, 2 weeks and 3 weeks. Clinical parameters were assessed at baseline and 6 weeks after root planing. Subgingival plaque was assessed at baseline and 6 weeks after root planing. Quantitative real-time PCR for Porphyromonas gingivalis (Pg), Treponema denticola (Td), Fusobacterium nucleatum (Fn) Tannerella forsythia (Tf) were performed at the same time.

SUMMARY:
Background: Chronic periodontitis is one of the most common causes of tooth loss and is rather common in the population. Treating chronic periodontitis remains a challenge for dental practitioners. The purpose of this study was to assess the clinical effects of sub-gingival application of 0.2% hyaluronic acid gel after root planing in the treatment of chronic periodontitis.

Materials and Methods: In this split mouth study, 733 periodontal pockets of 28 patients with moderate to severe chronic periodontitis were chosen for investigation. They were divided into 2 groups: control group and experimental group. The experimental group received sub-gingival administration of 1 ml of 0.2% hyaluronic acid gel into each pocket immediately after root planing and then after 1 week, 2 weeks and 3 weeks. Clinical parameters were assessed at baseline and 6 weeks after root planing. Subgingival plaque was assessed at baseline and 6 weeks after root planing. Quantitative real-time PCR for Porphyromonas gingivalis (Pg), Treponema denticola (Td), Fusobacterium nucleatum (Fn) Tannerella forsythia (Tf) were performed at the same time.

DETAILED DESCRIPTION:
Chronic periodontitis is one of the most common causes of tooth loss and is rather common in the population. Treating chronic periodontitis remains a challenge for dental practitioners. There are new applications of materials to promote the healing process and increase the effectiveness of treatment of CP such as antimicrobial and healing support agents which were used at scaling and root planing (SRP) phase with the desire to improve the effectiveness of treatment and reduce the frequency of surgical phase, in order to reduce treatment cost for patients. One of those materials is hyaluronic acid (HA).

HA is a polysaccharide with many important roles: maintaining stability, adjusting the viscosity of biological fluids, homeostasis, adjusting osmotic pressure, supporting structures ... The wide application of HA in medicine is due to its capability of binding multiple water molecules, bimproving tissue hydration and preventing mechanical damage, bacteriostatic, anti-inflamatory, osteoinductive.

This study was the first to be conducted in Vietnam to evaluate the effect of HA on the response of periodontal tissue in chronic periodontitis and its bactericidal efficiency. The bacteria we study were Porphyromonas gingivalis (Pg), Treponema denticola (Td), Fusobacterium nucleatum (Fn) Tannerella forsythia (Tf), which were important species in periodontitis development. The research results can supplement scientific evidence about the effects of this compound and clarify the usefulness of HA in clinical chronic periodontitis treatment.

We performed a randomized, controlled clinical trial with split-mouth design. Study procedure consisted of information collecting, clinical measurements and, data analysis. The study was conducted in full accordance with the World Medical Association Declaration of Helsinki 2000 and was registered at ClinicalTrials.gov No. 312/ĐHYD-HĐĐĐ.

Participants from 18 years old with a minimum number of 20 teeth who came for periodontitis treatment, were recruited at the Department of Periodontology, Faculty of Odonto-Stomalogy, the University of Medicine and Pharmacy at Ho Chi Minh City (FOS-UMPH). We selected patients with at least 3 teeth in the contralateral quadrants diagnosed with moderate or severe chronic periodontitis according to AAP (2015): gingival bleeding at examination, ≥5mm periodontal pocket depth, bone resorption on X-ray film ≥16% or >3mm root length.

Patients who were allergic to ingredients, being pregnant/lactating, smoking, alcoholic; who had undergone periodontal therapy in the last 6 months, received antibiotic therapy, anti-inflammatory agents, statins, drug induced gingival enlargement (such as phenytoin, cyclosporin, nifedipine) in the last 3 months were excluded. We also excluded patients with systemic diseases such as cardiovascular disease, hypertension, diabetes mellitus, or orthodontic treatment and patients who refused to participate in the study and/or follow-up visits.

According to Rajan (2014), to obtain the difference of probing pocket depth (PPD) of 2 groups (control and HA), we got and were the average PPD and 1.38 and were standard deviation of two groups, respectively. With α = 0.05 and β = 0.2, we calculated N = 25. 28 subjects were enrolled to prevent sample loss.

Masking of control and HA treatment were applied to patients, the periodontist and outcome assessing investigators for all clinical and laboratory parameters. Only an independent investigator who applied HA knew the name of the drug due to the nature of the study. Another investigator who performed the statistical assignment phase was to all patient information and to the following analysis and evaluation of the data.

In this split mouth study, 733 periodontal pockets of 28 patients with moderate to severe chronic periodontitis were chosen for investigation. They were divided into 2 groups: control group and experimental group. The experimental group received sub-gingival administration of 1 ml of 0.2% hyaluronic acid gel into each pocket immediately after root planing and then after 1 week, 2 weeks and 3 weeks. Clinical parameters were assessed at baseline and 6 weeks after root planing. Subgingival plaque was assessed at baseline and 6 weeks after root planing. Quantitative real-time PCR for Porphyromonas gingivalis (Pg), Treponema denticola (Td), Fusobacterium nucleatum (Fn) Tannerella forsythia (Tf) were performed at the same time. Wilcoxon sign-rank test and Mann-Whitney test were used for comparison of means.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 3 teeth in the contralateral quadrants diagnosed with moderate or severe chronic periodontitis according to AAP (2015): gingival bleeding at examination, ≥5mm periodontal pocket depth, bone resorption on X-ray film ≥16% or >3mm root length.

Exclusion Criteria:

* Patients who were allergic to ingredients, being pregnant/lactating, smoking, alcoholic; who had undergone periodontal therapy in the last 6 months, received antibiotic therapy, anti-inflammatory agents, statins, drug induced gingival enlargement (such as phenytoin, cyclosporin, nifedipine) in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | 6 weeks
  Periodontal pocket depth was evaluated at six positions in all teeth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual). The value of PPD was calculated by the total score/the number of positions.
Plaque index (PlI) | 6 weeks
  Plaque index (PlI) was evaluated at six positions in all teeth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual). The value of PlI was calculated by the total score/the number of positions.
Gingival index (GI) | 6 weeks
  Gingival index (GI) was evaluated at six positions in all teeth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual). The value of GI was calculated by the total score/the number of positions.
Clinical attachment loss (CAL) | 6 weeks
  Clinical attachment loss (CAL) was evaluated at six positions in all teeth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual). The value of CAL was calculated by the total score/the number of positions.
Bleeding on probing (BOP) | 6 weeks
  BOP was presented by the percentage of recorded bleeding sites.
Copy number of Porphyromonas gingivalis (Pg) | 6 weeks
  The copy number of Porphyromonas gingivalis (Pg) was monitored by Real-time PCR
Copy number of Treponema denticola (Td) | 6 weeks
  The copy number of Treponema denticola (Td) was monitored by Real-time PCR
Copy number of Fusobacterium nucleatum (Fn) | 6 weeks
  The copy number of Fusobacterium nucleatum (Fn) was monitored by Real-time PCR
Copy number of Tannerella forsythia (Tf) | 6 weeks
  The copy number of Tannerella forsythia (Tf) was monitored by Real-time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Thuy T Nguyen, PhD, Study Director — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Faculty of Odontostomatology - University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Shammari NM, Shafshak SM, Ali MS. Effect of 0.8% Hyaluronic Acid in Conventional Treatment of Moderate to Severe Chronic Periodontitis. J Contemp Dent Pract. 2018 May 1;19(5):527-534. PMID 29807962
- [Background] American Academy of Periodontology Task Force Report on the Update to the 1999 Classification of Periodontal Diseases and Conditions. J Periodontol. 2015 Jul;86(7):835-8. doi: 10.1902/jop.2015.157001. Epub 2015 May 27. No abstract available. PMID 26125117
- [Background] Bertl K, Bruckmann C, Isberg PE, Klinge B, Gotfredsen K, Stavropoulos A. Hyaluronan in non-surgical and surgical periodontal therapy: a systematic review. J Clin Periodontol. 2015 Mar;42(3):236-46. doi: 10.1111/jcpe.12371. Epub 2015 Mar 9. PMID 25640222
- [Background] Casale M, Moffa A, Vella P, Sabatino L, Capuano F, Salvinelli B, Lopez MA, Carinci F, Salvinelli F. Hyaluronic acid: Perspectives in dentistry. A systematic review. Int J Immunopathol Pharmacol. 2016 Dec;29(4):572-582. doi: 10.1177/0394632016652906. Epub 2016 Jun 8. PMID 27280412
- [Background] Eliezer M, Imber JC, Sculean A, Pandis N, Teich S. Hyaluronic acid as adjunctive to non-surgical and surgical periodontal therapy: a systematic review and meta-analysis. Clin Oral Investig. 2019 Sep;23(9):3423-3435. doi: 10.1007/s00784-019-03012-w. Epub 2019 Jul 23. PMID 31338632
- [Background] Gohler A, Hetzer A, Holtfreter B, Geisel MH, Schmidt CO, Steinmetz I, Kocher T. Quantitative molecular detection of putative periodontal pathogens in clinically healthy and periodontally diseased subjects. PLoS One. 2014 Jul 16;9(7):e99244. doi: 10.1371/journal.pone.0099244. eCollection 2014. PMID 25029268
- [Background] Rafiei M, Kiani F, Sayehmiri F, Sayehmiri K, Sheikhi A, Zamanian Azodi M. Study of Porphyromonas gingivalis in periodontal diseases: A systematic review and meta-analysis. Med J Islam Repub Iran. 2017 Sep 12;31:62. doi: 10.18869/mjiri.31.62. eCollection 2017. PMID 29445691
- [Background] Van der Weijden GAF, Dekkers GJ, Slot DE. Success of non-surgical periodontal therapy in adult periodontitis patients: A retrospective analysis. Int J Dent Hyg. 2019 Nov;17(4):309-317. doi: 10.1111/idh.12399. Epub 2019 May 16. PMID 30942938